CLINICAL TRIAL: NCT03822286
Title: E-training and Mentoring Support Program on Dementia Care for Home-care Workers
Brief Title: Development and Evaluation of E-training and Mentoring Support Program on Dementia Care for Home-care Workers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tzu Chi University (Other)
Responsible Party: Principal Investigator, Hsin Feng SU, Principal Investigator, Tzu Chi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: YLH-10721
Record Dates: First submitted 2019-01-27; First posted 2019-01-30 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Dementia
Keywords: home-care worker; e-training; mentoring support
MeSH Terms: conditions — Dementia | interventions — Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): E-training course programs, counseling mentoring supports and support group gatherings meeting.
  Interventions: Other: e-training course; Other: Support group
- Control (Active Comparator): Traditional classroom teaching course programs.
  Interventions: Other: traditional classroom teaching course programs

INTERVENTIONS:
Other: e-training course — Home care staff received mainly self-study, you can download e-books on your lithography or personal mobile phone reading and learning, with lively animation, sound and video guide home staff Learn the knowledge of demented care. The e-book course sets out the themes of the eight demented care training courses.
  Arms: Intervention
Other: Support group — A counseling master mix 8~10 resident staff members, through the counselor to lead the symposium to the case home to implement technical guidance and through the set of social network groups to immediately discuss the care and solutions of dementia cases, and hold once a month in gathering, about 40~60 minutes each time.
  Arms: Intervention
Other: traditional classroom teaching course programs — Home care staff received the traditional demented care traditional classroom teaching course and did not accept any e-training and gathering.
  Arms: Control

SUMMARY:
This study evaluate the effects of three-month dementia care e-training and mentoring support program on home-care workers using a two-group randomized controlled trial.

DETAILED DESCRIPTION:
Home care staff often have insufficient knowledge and skills of caring people with dementia at home. Many training courses for home care staff are not developed according to their educational background and workplace needs.

An innovative evidence-based online training with peer support program in dementia care was developed and consists of online cloud platform with various training courses and resources, on-the-job mentoring support by senior peers, and social networking in dementia care.

They can access to the online cloud platform by computers or smart phones anytime for immediate access to information in dementia care. They can also consult with senior peers for care problems by social network platform and attend monthly dementia care forum.

The interventional group attendance staff will accept 3-month e-training care online course, which was supervised by the supervisor and participated in the monthly counseling mentoring support group. The control group will accept the traditional dementedness care traditional classroom teaching course and will not accept any e-training .

The curriculum and counseling support group will collect information on the knowledge, attitudes, care abilities, work stress and burnout of the two groups in the pre-test, 3rd and 6th months and learn about their effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Qualified as a care worker for the elderly welfare law, and at least three months as a home servant,
* Literacy
* Can communicate in Mandarin and Taiwanese,
* Caring for community clients with cognitive impairment or dementia
* Willing to participate in the study and provide informed consent

Exclusion Criteria:

* If it does not meet the conditions for receiving the case, it will not be included in the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Dementia Knowledge Assessment Scale | 6 month
  To evaluate the staff care for knowledge of patients with dementia, range from 0-50, higher values represent the higher the care knowledge.
Approach to Dementia Questionnaire | 6 month
  To evaluate the staff care for Dementia care attitude, range from 19-95, higher values represent the more positive the attitude of the caregiver to dementia care.
Sense of Competence in Dementia Care Staff scale | 6 month
  To evaluate the staff care for demented patients, range from 16-68, higher values represent Staff have good care ability.
Maslach Burnout Inventory | 6 month
  To evaluate the Maslach Burnout Inventory,, range from 0-72, higher values represent a worse outcome.
Taiwan Simple Work Stress Scale | 6 month
  The main purpose is to measure the working pressure situation. The scale has a total of 38 questions, eight faces, each facing the score range of 0-100 points. The higher the score, the greater the work pressure.

CONTACTS AND LOCATIONS:
Overall Officials: HsinFeng SU, MSN, Principal Investigator — Tzu Chi University
Locations (1):
- HsinFeng,Su, Hualien City, Taiwan

REFERENCES:
- [Derived] Su HF, Koo M, Lee WL, Sung HC, Lee RP, Liu WI. A dementia care training using mobile e-learning with mentoring support for home care workers: a controlled study. BMC Geriatr. 2021 Feb 16;21(1):126. doi: 10.1186/s12877-021-02075-3. PMID 33593287